CLINICAL TRIAL: NCT06549595
Title: A Phase III, Multicentre, Randomised, Open-label Study to Compare the Efficacy and Safety of AZD0486 Plus Rituximab Versus Chemotherapy Plus Rituximab in Previously Untreated Participants With Follicular Lymphoma (SOUNDTRACK-F1)
Brief Title: A Study of Surovatamig (AZD0486) Plus Rituximab in Previously Untreated Follicular Lymphoma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7401C00001; 2023-510098-33-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Untreated Follicular Lymphoma
Keywords: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rituximab, Surovatamig - A (Experimental): Surovatamig regimen A plus rituximab
  Interventions: Drug: Surovatamig
- Rituximab, Surovatamig - B (Experimental): Surovatamig regimen B plus rituximab
  Interventions: Drug: Surovatamig
- Chemoimmunotherapy (Active Comparator): Investigator's choice between 3 standard immunochemotherapy regimen (R-CHOP, R-CVP, or B-R followed by rituximab maintenance)
  Interventions: Drug: R-CHOP; Drug: R-CVP; Drug: BR

INTERVENTIONS:
Drug: Surovatamig — a fully human bispecific monoclonal IgG4 antibody
  Other Names: AZD0486
  Arms: Rituximab, Surovatamig - A; Rituximab, Surovatamig - B
Drug: R-CHOP — Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone
  Arms: Chemoimmunotherapy
Drug: R-CVP — Rituximab, Cyclophosphamide, Vincristine and Prednisone
  Arms: Chemoimmunotherapy
Drug: BR — Bendamustine, Rituximab
  Arms: Chemoimmunotherapy

SUMMARY:
This is a global, randomised, Phase III, multicentre, open-label study evaluating the efficacy, safety and the degree of added benefit of the Surovatamig (AZD0486) plus rituximab combination compared to Investigator's choice of 3 standard immunochemotherapy regimen, conducted in participants with untreated FL.

DETAILED DESCRIPTION:
The study consists of 2 sequential parts.

1. Safety Run-in - this part will compare dose levels of Surovatamig (AZD0486) in combination with rituximab in order to establish the RP3D.
2. Phase III - The Phase III part will assess the superiority of Surovatamig (AZD0486) at RP3D in combination with rituximab, compared to Investigator's choice between 3 standard chemoimmunotherapy regimens. Phase 3 consists of 3 arms

   1. Arm A: treatment with Surovatamig plus rituximab Schedule A
   2. Arm B: treatment with Surovatamig plus rituximab Schedule B
   3. Arm C (Comparator arm): one of the following standard regimens per Investigator's choice: R-CVP + rituximab maintenance, R-CHOP + rituximab maintenance or B-R + rituximab maintenance

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age, inclusive, at the time of signing the ICF.
2. Histologically confirmed diagnosis of classic FL per WHO 2022 classification
3. ECOG performance status of 0 to 2
4. No prior systemic lymphoma-directed therapy
5. Need for systemic treatment meeting at least 1 GELF criteria
6. FDG-avid and measurable disease
7. Stage II to IV and FLIPI 2-5 [Phase III only]
8. Adequate liver, hematological, renal and cardiac function.

The above is a summary, other inclusion criteria details may apply

Exclusion Criteria:

1. Follicular large B-cell lymphoma (WHO 2022 classification), formerly Follicular lymphoma Grade 3B (WHO 2016 classification) or suspicion for histologic transformation to high-grade/aggressive lymphoma
2. Contra-indication to BR, RCVP, and R-CHOP
3. Participants with or history of CNS lymphoma
4. History of a clinically relevant CNS medical condition or pathology that required treatment in the preceding year, is currently symptomatic or that which the treating investigator considers to have the potential to interfere with the evaluation of safety
5. Presence of >5000 circulating lymphoma cells
6. Active or uncontrolled infection (including EBV) requiring systemic therapy and which places participant at unacceptable risk if he/she were to participate in the study. If a participant has a history of COVID-19 within 1 month of C1D1 or contracts COVID while on study treatment, participant must have 2 consecutive negative tests (PCR testing is preferable) performed at least 48 hours apart prior to resuming dosing. All symptoms related to COVID-19 infection should have fully resolved before initiating or resuming treatment
7. Known history of hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS)

The above is a summary, other exclusion criteria details may apply

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2031-11-26 (Estimated); Study Completion 2031-11-26 (Estimated)

PRIMARY OUTCOMES:
SRI Primary: Incidence, nature and severity of AEs and SAEs. Incidence and nature of study drug discontinuations, dose reductions, and dose delays due to AEs | Up to 10 years
  Frequency, severity, and relationship to study drug of AEs and SAEs; dose modifications; changes in physical examination and safety procedures.
SRI Primary: Determination of the recommended Phase III dose (RP3D) | Up to 1 year
  The RP3D will be the dose of Surovatamig selected for the Phase 3 part based on safety data compiled during the safety run-in part
Phase 3 Dual Primary: To demonstrate the superiority of Surovatamig plus rituximab compared to Investigator's choice of SoC chemoimmunotherapy | Up to 10 years
  PFS, based on Lugano 2014 Response Criteria, as assessed by BICR.
Phase 3 Dual Primary: To demonstrate the superiority of Surovatamig plus rituximab compared to Investigator's choice of SoC chemoimmunotherapy | Up to 10 years
  ORR at EoI, based on Lugano 2014 Response Criteria, as assessed by BICR.

SECONDARY OUTCOMES:
Safety Run in and Phase 3: ORR at EoI (Investigator assessed) | Up to 10 years
  ORR defined as the proportion of participants achieving either a PR or CR at End of Induction based on Lugano 2014 Response Criteria
Safety Run In and Phase 3: CR Rate | Up to 10 years
  CR rate is defined as the proportion of participants achieving a CR at any time as based on Lugano 2014 Response Criteria
Safety Run In and Phase 3: CR at EoI | Up to 10 years
  Proportion of participants achieving CR at End of Induction based on Lugano 2014 Response Criteria
Safety Run In and Phase 3: DoR | up to 10 years
  DoR will be defined from the time of first response until progression based on Lugano 2014 criteria, or death due to any cause
Safety Run In and Phase 3: PFS (Investigator assessed) | Up to 10 years
  PFS (Investigator assessed) is defined as time from randomization until disease progression based on Lugano 2014 Response Criteria or death due to any cause
Safety Run In and Phase 3: OS | Up to 10 years
  OS is defined as time until the date of death
Phase 3: CR rate at 30 months (CR30) | Up to 30 months
  Proportion of participants in CR rate at 30 months (CR30) based on Lugano 2014 Response Criteria
Phase 3: Time to First Subsequent Therapy or Death (TFST) | Up to 10 Years
  TFST will be defined as the time from randomization until the start date of first subsequent anti-lymphoma therapy or death due to any cause
Phase 3: Time from randomisation to second progression or death (PFS2) | Up to 10 Years
  PFS2 will be defined as the time from randomization until the earliest of the progression event, after first subsequent therapy, or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chan Cheah, MBBS FRACP FRCPA DMSc, Principal Investigator — Sir Charles Gairdner Hospital (SCGH)
Locations (104):
- Australia (4):
  - Research Site, Garran
  - Research Site, Heidelberg
  - Research Site, Macquarie University
  - Research Site, Nedlands
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Mechelen
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jérôme, Quebec
- China (25):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Tampere
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Research Site, Budapest, Hungary
- India (6):
  - Research Site, Delhi
  - Research Site, Gurugram
  - Research Site, Kolkata
  - Research Site, Nashik
  - Research Site, Surat
  - Research Site, Thiruvananthapuram
- Japan (18):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chuo-shi
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurashiki-shi
  - Research Site, Kyoto
  - Research Site, Minatoku
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Yamagata
  - Research Site, Yokohama
- Research Site, Gliwice, Poland
- South Korea (4):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Jeonnam
  - Research Site, Seoul
- Spain (8):
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Girona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santander
- Sweden (2):
  - Research Site, Falun
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Lukang Township
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
- Research Site, Ankara, Turkey (Türkiye)
- United Kingdom (6):
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home